CLINICAL TRIAL: NCT07049003
Title: Deep Brain Stimulation of the Deep Cerebellar Nuclei for Refractory Tremor
Acronym: rT DBS
Status: Recruiting | Phase: Phase 1 | Type: Interventional
Sponsor: The Cleveland Clinic (Other)
Collaborators: Raynor Cerebellum Project (Unknown); Medtronic (Industry)
Responsible Party: Principal Investigator, Andre Machado, Institute Chief Neurological Institute, The Cleveland Clinic
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 25-182
Record Dates: First submitted 2025-05-28; First posted 2025-07-03 (Actual); Last update posted 2025-07-03 (Actual); Status verified 2025-06

CONDITIONS: Tremor; Essential Tremor
MeSH Terms: conditions — Tremor; Essential Tremor | interventions — Deep Brain Stimulation

STUDY DESIGN:
Intervention Model Description: All subjects will receive open label deep brain stimulation implantation of the deep cerebellar nuclei
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: Yes

ARMS (1):
- Refractory Tremor (Experimental): Medtronic Percept RC DBS System
  Interventions: Device: Deep Brain Stimulation

INTERVENTIONS:
Device: Deep Brain Stimulation — Deep Brain Stimulation of the Deep Cerebellar Nuclei
  Other Names: Medtronic Percept DBS System

SUMMARY:
This objective of this study is to document the safety and feasibility of electrical stimulation of the deep cerebellar nuclei for refractory tremor using the Medtronic Percept RC Deep Brain Stimulation System. The population will consist of patients that have either failed a prior intervention (Vim DBS or HIFU thalamotomy) or determined to not be suitable candidates for Vim DBS or HIFU thalamotomy because they have a cerebellar outflow or MS-related tremor. Those patients with a previous intervention, must have a prior diagnosis of ET, cerebellar outflow tremor, or MS-related tremor. Subjects without a previous intervention must have a diagnosis of cerebellar outflow tremor or MS-related tremor.

ELIGIBILITY:
Inclusion Criteria:

* Age 21 years and older;
* Ability to give informed consent;
* Diagnosis of ET, cerebellar tremor, or MS-related tremor with a failed a prior intervention (VIM DBS or HIFU thalamotomy) or determined to not be suitable candidates for VIM DBS or HIFU thalamotomy because they have a cerebellar outflow or MS-related tremor.
* Tremor history of at least three years;
* Tremor that is refractory to medical management;
* A score of ≥24 on the Mini Mental State Examination;
* Inability to successfully perform ADLs without assistance or has lost interest in social, professional, or personal activities due to tremor

Exclusion Criteria:

* Any other neurological condition that could reduce the safety of study participation including central nervous system vasculitis and intracranial malignancy
* A condition that, in the opinion of the clinical investigator, would significantly increase the risk or interfere with study compliance, safety, or outcome;
* A diagnosis of dementia;
* Tremors due to other neurological conditions such as Parkinson's disease, dystonia, or other conditions not consistent with ET, cerebellar outflow tremor, or MS-related tremor.
* Diagnosis of epilepsy;
* Major active and untreated psychiatric illness that may interfere with study, such as psychotic disorders or severe personality disorders;
* Untreated or inadequately treated depression defined by a score of 20 or greater on the Beck Depression Inventory-II at the time of enrollment;
* At risk for suicide defined by a score greater or equal to 3 on the Columbia Suicide Severity Rating Scale (C-SSRS);
* Pregnancy;
* Unable to communicate with investigators or staff;
* Surgical contraindications to DN DBS;
* Contraindication to magnetic resonance (MRI) imaging, e.g., weight incompatible with scanner, implanted metallic devices or electrical devices (pacemaker, defibrillator, spinal cord stimulator, prior DBS) or intolerance to MRI contrast agent;
* Enrolled in another device, biologic or pharmaceutical study within 30 days of consent in the current study, (i.e., patient cannot be enrolled if participation in another study was not completed at least 30 days prior to consent.);
* Evidence of behavior(s) consistent with alcohol or substance abuse/dependence as defined by the criteria outlined in the DSM-V within the preceding six months;
* Injection of botulinum toxins into the arm, neck or face within six months prior to baseline;

Min Age: 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 12 (Estimated)
Dates: Start 2025-05-19 (Actual); Primary Completion 2028-12-31 (Estimated); Study Completion 2028-12-31 (Estimated)

PRIMARY OUTCOMES:
The incidence and nature of treatment-related adverse events | From DBS Implant Surgery through study completion, an average of 17 months
  The accumulation of adverse events across all subjects

SECONDARY OUTCOMES:
Fahn Tolosa Marin Tremor Rating Scale | From DBS Implant Surgery through study completion, an average of 17 months
  An objective measurement of the severity of tremor. A 32-part questionnaire that evaluates tremor severity by assigning a numerical value of 0-4 to the answers for 32 questions. Numerical values are added together for a total score. A higher score represents a more severe tremor than a lower score.
DBS-evoked potentials | From DBS Implant Surgery through study completion, an average of 17 months
  The prevalence and strength of markers of electrophysiological activity across the cerebellothalamocorticomuscular (CTCM) network at rest and during tremor-eliciting motor behaviors.
4-8 HZ (theta) tremor related oscillations | From DBS Implant Surgery through study completion, an average of 17 months
  Examination of how the DN and VIM DBS (when present) modulate oscillatory activity and coupling across the CTCM circuit in relation to improvements in tremor control. A 4-8Hz (theta) tremor-related oscillation is observed consistently in the VIM during motor activity, which parallels the activity-dependent appearance of tremor in patients with ET.

CONTACTS AND LOCATIONS:
Locations (1):
- Cleveland Clinic, Cleveland, Ohio, United States

IPD SHARING:
Plan to Share IPD: No